CLINICAL TRIAL: NCT01799434
Title: Influence of an Exercise on the Dynamic Postural Control in Athletes
Brief Title: Dynamic Postural Control After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. med. Benita Kuni, MD, Specialist for Orthopedics and Trauma Surgery, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 407-05-130203
Record Dates: First submitted 2013-02-19; First posted 2013-02-26 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Postural Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): All participants had to run 20min on their individual anaerobic threshold
  Interventions: Other: treadmill run

INTERVENTIONS:
Other: treadmill run

SUMMARY:
The aim was to analyze the influence of fatigue on the dynamic postural control in one-leg standing and in jump landing, followed by stabilization or side jumps, and to compare athletes of different levels with control subjects.

ELIGIBILITY:
Inclusion Criteria:

* competitive level (participation in any league) for the high performance athletes group
* participation in sport for 0.5-4 hours per week for the recreationally active subjects

Exclusion Criteria:

* current history of a lower extremity injury requiring training cessation on the day of testing
* neurological diseases
* vestibular or visual disturbances
* cardiovascular diseases medication affecting balance

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change of force ratio of ground reaction forces in/after landing from baseline | 1, 5, 10, 15, 20 min after exercise
Change of the velocity of the center of pressure (COP) from baseline | 1, 5, 10, 15, 20 min after the exercise

SECONDARY OUTCOMES:
Change of rate of perceived exertion (Borg Scale) from baseline | every 10 min during and 1, 5, 10, 15, 20 min after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Department of Orthopedics, Trauma Surgery and Spinal Cord Injury, Heidelberg, Germany